CLINICAL TRIAL: NCT06739694
Title: The Efficacy of a Pain Neuroscience Education Programme in Shoulder Pain: a Randomised Clinical Trial
Brief Title: Neuroscience Education in Shoulder Pain: Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Eva Prado Robles, Principal Investigator and clinical Professor, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SALUD DOCTORADO
Record Dates: First submitted 2024-12-08; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Shoulder Pain
Keywords: exercise; manual therapy; shoulder pain; pain neuroscience education
MeSH Terms: conditions — Shoulder Pain; Motor Activity | interventions — Musculoskeletal Manipulations; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Participants will receive 4 sessions of PNE and 5 sessions of manual therapy and exercises.
  Interventions: Behavioral: PNE; Procedure: Manual therapy
- Control group (Active Comparator): Participants will receive 5 sessions of manual therapy and exercises.
  Interventions: Procedure: Manual therapy

INTERVENTIONS:
Behavioral: PNE — A manual therapy(Mulligan´s Mobilization with Movement) and 4 sessions of strenght exercises program was administered for both groups. In addition, a pain neuroscience education protocol was administered for the experimental group for a whole period of 4 weeks (1 session/week, 75mins per session).
  Other Names: Manual therapy; Exercise
  Arms: Experimental group
Procedure: Manual therapy — 5 sessions of Mulligan´s Mobilization with Movement and 4 sessions of strenght exercises

SUMMARY:
Objectives: The purpose of this study was to assess the efficacy of a pain neuroscience education programme applied to patients with shoulder pain.

DETAILED DESCRIPTION:
A randomised controlled trial was performed. Fifty-five patients satisfied eligibility criteria, agreed to participate, and were randomized into an experimental group (n = 27) or control group (n =28). A manual therapy and exercises program was administered for both groups. In addition, a pain neuroscience education protocol was administered for the experimental group for a whole period of 4 weeks (1 session/week, 75mins per session).

ELIGIBILITY:
Inclusion Criteria:

* Being 18-70 years of age.
* History of shoulder pain of more than 3 months duration.
* Presence of a painful arc
* Medical diagnosis of shoulder pain with at least 2 positive impingement tests including Neer, Hawkins, or Jobe test

Exclusion Criteria:

* Diagnosis of fibromyalgia.
* Pregnancy.
* A history of traumatic onset of shoulder pain.
* Other histories of shoulder injury.
* Torn tendons.
* Ligamentous laxity based on a positive Sulcus and apprehension tests.
* Numbness or tingling in the upper extremity.
* Previous shoulder or cervical spine surgery.
* Systemic illness.
* Corticosteroid injection on the shoulder within 1 year of the study.
* Physical therapy 6 months before the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Pain | Baseline and 5 weeks.
  Reduction in pain intensity using the Shoulder Pain and Disability Index (SPADI)
Disability | Baseline and five weeks.
  Improving functionality using the Shoulder Pain and Disability Index (SPADI)

SECONDARY OUTCOMES:
kinesiophobia | Baseline and 5 weeks.
  Tampa Scale of Kinesiophobia (TSK11)

OTHER OUTCOMES:
catastrophizing | Baseline and 5 weeks.
  Pain catastrophizing scale (PCS)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Prado Robles, Principal Investigator — Universidad de León
Locations (1):
- Eva, León, Spain, Spain

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared due to ethical and legal restrictions on the privacy of participants.

REFERENCES:
- [Background] Wood L, Hendrick PA. A systematic review and meta-analysis of pain neuroscience education for chronic low back pain: Short-and long-term outcomes of pain and disability. Eur J Pain. 2019 Feb;23(2):234-249. doi: 10.1002/ejp.1314. Epub 2018 Oct 14. PMID 30178503